CLINICAL TRIAL: NCT03218930
Title: Maltese Antibiotic Stewardship Programme in the Community (MASPIC): a Prospective Quasi-experimental Social Marketing Intervention
Brief Title: Maltese Antibiotic Stewardship Programme in the Community (MASPIC): Antibiotic Prescribing for Acute Respiratory Tract Complaints
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: University of Malta (Other)
Responsible Party: Principal Investigator, Erika Saliba Gustafsson, Doctoral student, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MASPIC
Record Dates: First submitted 2017-07-10; First posted 2017-07-17 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Acute Respiratory Infection
Keywords: General Practice; Social Marketing; Behavior Change; Antibiotic Prescribing
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social marketing intervention (Other): Participants will receive a total combination of four interventions.
  Interventions: Behavioral: Delayed antibiotic prescription; Behavioral: Antibiotic prescribing guidelines; Behavioral: Education; Behavioral: Educational materials

INTERVENTIONS:
Behavioral: Delayed antibiotic prescription — Delayed antibiotic prescription pads will be disseminated to all participating general practitioners in both hard and soft copies.
Behavioral: Antibiotic prescribing guidelines — Antibiotic prescribing guidelines will be disseminated to all participating general practitioners in both hard and soft copies.
Behavioral: Education — General practitioners will receive a package of educational sessions tailored towards their specific needs.
Behavioral: Educational materials — Educational materials for patients, namely posters and leaflets, will be disseminated to all participating general practitioners.

SUMMARY:
Antibiotic resistance has become a major threat to global public health. It is driven by a multitude of factors, however one of the leading factors is antibiotic prescribing. Inappropriate antibiotic use and overuse of broad-spectrum antibiotics can lead to the development of resistant strains. Since in Malta the vast majority of antibiotics are acquired through prescription, targeting providers' prescribing behavior is an important strategy needed to try to curb antibiotic overuse and resistance.

The aim of this study is to evaluate the effect of a multifaceted social marketing intervention in changing general practitioners' (GPs) antibiotic prescribing behavior for patients with acute respiratory tract complaints in Malta. This quasi-experimental intervention study using an interrupted time series design includes three phases; a formative pre-intervention phase, an intervention phase and post-intervention evaluation phase, and will last a total of four years.

During the pre-intervention phase, various stakeholders, including GPs, pharmacists and parents will be interviewed in order to get a better contextual understanding of antibiotic use in Malta. A 1-year baseline surveillance system will also be set up to collect actual diagnosis-specific antibiotic prescribing by GP. This data will, at a later stage, be used to measure the change in antibiotic prescribing behavior post-intervention stage. GPs stage of behavior change and intention to prescribe antibiotics will also be measure pre-intervention using questionnaires based on the theory of planned behavior and the transtheoretical model.

The intervention stage will last 6 months and will include multiple components, including, delayed prescription pads, educational sessions, educational materials for patients and distribution of antibiotic guidelines. The intervention will be monitored closely through numerous process indicators.

Following the intervention, GPs' stage of change and intention to prescribe antibiotics will be re-measured using the same questionnaire used pre-intervention. Surveillance data collection will be also be resumed and will provide data to measure the primary outcome as well as additional secondary outcomes.

The primary outcome of interest is the change in the rate of antibiotic prescribing for patients presenting with an acute respiratory tract complaint.

ELIGIBILITY:
Inclusion Criteria:

* All actively practicing general practitioners and trainees specializing within family medicine are eligible to participate regardless of whether they work on a part-time or full-time basis, or in the public and/or private sectors

Exclusion Criteria:

* General practitioners who are no longer actively working

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
The antibiotic prescribing rate for patients with acute respiratory tract complaints. | Three years
  An interrupted time series design will allow us to measure the change in the antibiotic prescribing rate post-intervention compared with the pre-intervention phase through segmented regression analysis. Surveillance data will be collected pre- and post-intervention using a tool adapted from previous research. The tool will be piloted locally and checked for face validity.

SECONDARY OUTCOMES:
The proportion of diagnosis-specific antibiotic prescription, specifically for the common cold, acute pharyngitis, acute sinusitis, acute bronchitis, acute tonsillitis, acute otitis media, pneumonia, allergy and influenza | Three years
  The change in diagnosis-specific antibiotic prescribing rates post-intervention compared with the pre-intervention phase will be analysed using segmented regression.
The proportion of symptomatic relief medication prescribed | Three years
  The change in the proportion of symptomatic relief medication prescribed post-intervention compared with the pre-intervention phase will be analysed.
The change in general practitioners' (GPs) stage-of-change | Three years
  In order to be able to measure the change in GPs' stage of behavior change post-intervention, a questionnaire will be developed based on the transtheoretical model (or stage-of-change theory) and distributed to GPs pre- and post-intervention. The questionnaire will be informed by previous studies and adapted to the local context.
The change in general practitioners' (GPs) behavioral intention to prescribe antibiotics | Three years
  In order to be able to measure the change in GPs' intention to prescribe antibiotics post-intervention, a questionnaire will be developed based on the theory of planned behavior and distributed to GPs pre- and post-intervention. The questionnaire will be informed by previous studies and adapted to the local context.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Stålsby Lundborg, Prof, Principal Investigator — Karolinska Institutet

REFERENCES:
- [Derived] Saliba-Gustafsson EA, Nyberg A, Borg MA, Rosales-Klintz S, Stalsby Lundborg C. Barriers and facilitators to prudent antibiotic prescribing for acute respiratory tract infections: A qualitative study with general practitioners in Malta. PLoS One. 2021 Feb 11;16(2):e0246782. doi: 10.1371/journal.pone.0246782. eCollection 2021. PMID 33571265
- [Derived] Saliba-Gustafsson EA, Dunberger Hampton A, Zarb P, Orsini N, Borg MA, Stalsby Lundborg C. Factors associated with antibiotic prescribing in patients with acute respiratory tract complaints in Malta: a 1-year repeated cross-sectional surveillance study. BMJ Open. 2019 Dec 18;9(12):e032704. doi: 10.1136/bmjopen-2019-032704. PMID 31857311
- [Derived] Saliba-Gustafsson EA, Roing M, Borg MA, Rosales-Klintz S, Lundborg CS. General practitioners' perceptions of delayed antibiotic prescription for respiratory tract infections: A phenomenographic study. PLoS One. 2019 Nov 22;14(11):e0225506. doi: 10.1371/journal.pone.0225506. eCollection 2019. PMID 31756197
- [Derived] Saliba-Gustafsson EA, Borg MA, Rosales-Klintz S, Nyberg A, StalsbyLundborg C. Maltese Antibiotic Stewardship Programme in the Community (MASPIC): protocol of a prospective quasiexperimental social marketing intervention. BMJ Open. 2017 Sep 24;7(9):e017992. doi: 10.1136/bmjopen-2017-017992. PMID 28947463